CLINICAL TRIAL: NCT05867953
Title: A Prospective Investigation to Assess the Accurate Tool Placement in Pulmonary Nodule(s) Using a Robotic Navigational Bronchoscopy System With Adjunct Real-time Imaging
Brief Title: Assessment of Tool Placement in Pulmonary Nodule(s) Using a Robotic Navigational Bronchoscopy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISI-ION-EU1-2022
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Biopsy; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, single-arm, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biopsy Arm (Experimental): Patients undergoing biopsy with the Ion Endoluminal System
  Interventions: Device: Biopsy with the Robotic- Ion Endoluminal System with Adjunct Real-time Imaging

INTERVENTIONS:
Device: Biopsy with the Robotic- Ion Endoluminal System with Adjunct Real-time Imaging — Biopsy with the Robotic- Navigational Bronchoscopy System with Adjunct Real-time Imaging

SUMMARY:
The aim of this research study is to evaluate the effectiveness of the ION endoluminal system at reaching and obtaining biopsies from lung nodules when used in combination with 3-dimensional imaging such as CT scans. Data on safety will also be collected.

DETAILED DESCRIPTION:
This is a prospective, interventional, multicentre, single arm study which will be conducted in Europe and will involve up to 200 patients undergoing a pulmonary nodule biopsy using the Ion Endoluminal System in conjunction with 3D imaging.

The objectives of the study are focused on evaluating the procedure characteristics of the pulmonary nodule biopsy procedure, including rate of tool in nodule, diagnostic accuracy, sensitivity for malignancy and safety.

All subjects will be followed up at 1 week and 1 month after the procedure. If the biopsy did not provide a diagnosis or did not show cancer and was still under observation at the 1 month visit, then they will have further follow up at 6 months. Similarly, if the status is unchanged (non-malignant diagnosis) at 6 months, the patients a 13 months visit should be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 18 years or older at time of consent.
2. Patient is suitable for elective nodule biopsy via bronchoscopy under general anesthesia per Investigator's discretion.
3. Patient has solid or semi-solid pulmonary nodule(s) of ≥6 mm and ≤3 cm in largest dimension (based on pre-procedure CT scan).
4. Pulmonary nodule(s) intended for biopsy during the study procedure is (are) located at least 4 (≥4) airway generations out (trachea = generation 0, e.g. subsegmental bronchi or beyond) based on pre-procedure CT scan.
5. Patient has a moderate to high risk of lung cancer based on clinical, demographic, and radiologic information or with suspected metastatic disease. High risk for malignancy patients are eligible if a biopsy is required or requested prior to intervention.
6. Patient is willing and able to give written informed consent for Clinical Investigation participation.
7. Patient is not legally incapacitated or in a legal/court ordered institution.

Exclusion Criteria:

1. Patient has a lack of fitness or exercise capacity to undergo bronchoscopy under general anesthesia as determined by Investigator prior to procedure.
2. Patient with type 1 pure ground glass opacity target nodule(s) intended for biopsy during study procedure.
3. Presence of mediastinal or hilar lymphadenopathy requiring tissue biopsy on pre-procedure CT or positron emission tomography (PET)-CT scan.
4. Patient with American Society of Anesthesiologists Classification (ASA) ≥4.
5. Patient underwent a pneumonectomy.
6. Any invasive concomitant procedure not related to the pulmonary nodule(s) or suspected disease state.
7. Female patient of child-bearing potential who is unable to take adequate contraceptive precautions or is known to be pregnant, and/or breast feeding.
8. Patient has a documented medical history of uncorrectable coagulopathy, bleeding, or platelet disorder.
9. Patient is taking antiplatelet or anticoagulant medications that cannot be stopped per standard practice.
10. Patient is currently participating or has participated in another Clinical Investigation within the past 30 days, such as interventional trials or trials with experimental agents or agents of unknown risk, that may affect the endpoints of this Clinical Investigation.
11. Investigator, in their professional opinion, has decided that it is in the patient's best interest to not participate in the Clinical Investigation.
12. Patient is not willing to comply with post study procedure participation requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Tool in Nodule | At time of the biopsy procedure (Day 0)
  Rate of achieving biopsy tool position within the targeted nodule(s), documented by means of intraprocedural 3D imaging.
  Defined as how often the biopsy needle used to sample the tissue is positioned directly within the nodule before the sample is taken.
  If biopsy forceps are used, it is how often the instrument is surrounding the nodule before the sample is taken

SECONDARY OUTCOMES:
Diagnostic accuracy of sample(s) obtained | Up to 13 months post procedure
  Diagnostic accuracy will be calculated as the rate of diagnosis made using samples obtained during the study procedure (true positives and true negatives) relative to the number of cases performed.
  Diagnostic yield may also be reported in conjunction with diagnostic accuracy and calculated as the rate of malignant and benign diagnosis made relative to the number of cases performed; non-diagnostic samples will not be included in the numerator.
Sensitivity for malignancy of sample(s) obtained | Up to 13 months post procedure
  Sensitivity for malignancy of samples is assessed as the number of subjects with a malignant condition determined through the study procedure (true positives) relative to the number of subjects with an underlying malignant disease state (true positives + false negatives). The subjects underlying disease state will be determined by follow-up diagnostic interventions or treatment decisions/interventions, and/or radiographic follow-up.

OTHER OUTCOMES:
Rate of procedure-related Adverse Events through 30 days post-procedure | 30 days
  The study's safety endpoint is the rate of procedure-related Adverse Events through 30 days post-procedure
Exploratory endpoint 1: Procedure-related characteristics | At time of the biopsy procedure (Day 0)
  Procedure time (from catheter inserted into the patient's airways to catheter removed from the patient's airways) will be reported.
Exploratory endpoint 2:rEBUS visualization characteristics | At time of the biopsy procedure (Day 0)
  The frequency of rEBUS visualization view during the biopsy will be summarized.
Exploratory endpoint 3: Biopsy workflow | At time of the biopsy procedure (Day 0)
  The sequence of biopsy tools used will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Master, Study Director — Intuitive Surgical
Locations (2):
- United Kingdom (2):
  - Barts Health Nhs Trust, London
  - Royal Brompton & Harefield Hospitals, Part of Guy'S and St Thomas' Nhs Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan LT, Lau KKW, Orton CM, Temov K, Tana A, Baboolal I, Karir A, Agaoglu E, Garner J, Kalyal A, Lapuente M, Ttofia F, Shah PL. Tool in lesion verification of shape-sensing robotic-assisted bronchoscopy with cone beam CT in sampling peripheral pulmonary nodules. Thorax. 2025 Dec 18:thorax-2025-223631. doi: 10.1136/thorax-2025-223631. Online ahead of print. PMID 41391887